CLINICAL TRIAL: NCT01156896
Title: Malaria and Iron Intervention Safety: Absorption and NTBI
Brief Title: Malaria and the Safety of Iron Supplements and Iron Fortification
Acronym: MIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gary M Brittenham, MD, James A Wolff Professor of Pediatrics, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAF0995; U01HD061233-04 (NIH)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Iron Deficiency
Keywords: Non-transferrin-bound iron; Iron stable isotopes; Iron deficiency; Malaria; Iron supplementation; Iron fortification
MeSH Terms: conditions — Iron Deficiencies; Malaria | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron intervention (Experimental): All study subjects with malaria and all control subjects will receive an iron intervention (supplement or fortification dose of iron).
  Control subjects will be studied on only one occasion.
  Study subjects with malaria will receive the same iron intervention two weeks later, after the malarial episode has been successfully treated.
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — Ferrous sulfate, ~1 mg Fe/kg body weight, given as a single dose in the fasting state.
Dietary Supplement: Ferrous sulfate — Ferrous sulfate, ~1 mg Fe/kg body weight, given as a single dose with a standard Thai rice meal.
Dietary Supplement: Ferrous sulfate — Ferrous sulfate, ~1 mg Fe/kg body weight, given as a single dose with a standard Thai rice meal with added oil.
Dietary Supplement: Ferrous sulfate — Ferrous sulfate, ~0.1 mg Fe/kg body weight, given as a single dose with a standard Thai rice meal.

SUMMARY:
The primary study hypothesis of the investigators is that administration of an iron supplement between meals at a dose like that used in the Pemba trial (~1 mg Fe/kg) during P. falciparum parasitemia will increase plasma non-transferrin-bound iron. A key subsidiary hypothesis is that iron administered with meals in amounts used in food fortification (~0.1 mg Fe/kg) will not produce plasma non-transferrin-bound iron.

This research will be carried out at the Hospital for Tropical Diseases, Mahidol University, Bangkok, Thailand. The studies are intended to help understand how giving iron and folic acid to preschool children in Pemba, Zanzibar, Tanzania, (the "Pemba trial") in the doses recommended by the World Health Organization, could have resulted in an increase in hospitalizations and deaths. The investigators will examine the most likely explanation, that the dose of iron supplements used in the Pemba trial produced iron in the blood not bound to the usual carrier for iron (a protein called "transferrin"), that is called "non-transferrin-bound iron", abbreviated as NTBI. In children with malaria, this NTBI might favor the growth of malarial parasites or other causes of infection. At present, no studies have been carried out to see if NTBI is present after giving iron to patients with malaria. Using non-radioactive forms of iron (called "stable isotopes"), the investigators will study iron absorption and NTBI after giving a single dose of iron (like that used in the Pemba trial) one day after treatment for malaria has been started, while patients still have malaria parasites in the blood, and then again two weeks later, after the malaria has been cured. The investigators will study adults admitted to the Hospital for Tropical Diseases in Bangkok, Thailand, with malaria. For reasons of safety, the investigators have chosen to study adults in the hospital rather than children living in an area like Pemba but the results should also apply to children. The outcome of this research will help us design ways of safely giving iron in malarious areas to adults and children to prevent or treat iron deficiency.

DETAILED DESCRIPTION:
This research will determine the effects of acute infection with Plasmodium falciparum on the absorption, pharmacokinetics and metabolism of iron from iron supplements and other iron preparations in non-immune adults in Thailand. Our project will combine measurements of iron absorption during and after successful treatment of acute uncomplicated falciparum malaria with characterization of the pharmacokinetics of the appearance of plasma nontransferrin-bound iron (NTBI) and measurements of the iron regulatory hormone, hepcidin, and other proteins of iron metabolism. We will examine iron supplements like those used in the Pemba supplementation trial (Sazawal et al., Lancet 2006; 367, 133-143) as well as alternative iron interventions that could minimize or avoid the formation of plasma non-transferrin-bound iron. This research has three specific aims:

1. to characterize the pharmacokinetics of the appearance of non-transferrin bound iron in the systemic circulation after oral administration of an iron supplement or other iron intervention;
2. to determine the effect of acute uncomplicated falciparum malaria on absorption of iron from iron supplements and other iron interventions, using erythrocyte incorporation of stable isotopes of iron;
3. to assess the effects of acute uncomplicated falciparum malaria on iron metabolism by repeated measurements of serum hepcidin, transferrin receptor, ferritin, haptoglobin, and concentrations of pro- (Th-1) and anti- (Th-2) inflammatory cytokines, erythrocyte zinc protoporphyrin, and the complete blood count with absolute reticulocyte count and reticulocyte hemoglobin content (CHr).

These studies of the effects of infection with P. falciparum on iron absorption and metabolism will further our basic understanding of the interaction of iron supplements with malaria and other infections. The results could help guide the choice of optimal means for the prevention and treatment of iron deficiency in regions endemic for malaria. Characterization of the pharmacokinetics of changes in plasma iron produced by administration of conventional iron supplements could lead to the design and development of new formulations of supplemental iron that would maximize iron absorption while minimizing risks associated with non-transferrin-bound plasma iron. Because of the public health importance of assuring iron sufficiency in mothers, our studies are focused on women of childbearing age but the results should be broadly applicable to the optimal means of providing iron to infants and children.

ELIGIBILITY:
Inclusion Criteria:

* men or premenopausal woman, 18 to 50 years of age;
* peripheral blood positive for asexual forms of P. falciparum (this criterion not applicable to uninfected healthy control subjects);
* women not pregnant by self-report and not planning pregnancy;
* body weight <65 kg.

Exclusion Criteria:

* presence of severe or complicated malaria as defined by WHO criteria;
* clinical evidence of ill health or a history of chronic disorders;
* treatment for mental illness;
* imprisonment;
* institutionalization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma non-transferrin-bound iron (NTBI) | 0, 2, 4, 8, 12 and 24 hours
  After administration of an iron intervention, plasma non-transferrin-bound iron pharmacokinetics will be determined.

SECONDARY OUTCOMES:
Erythrocyte 58Fe incorporation | Determined 2 weeks after iron intervention
  Erythrocyte 58Fe incorporation will be measured using stable-isotope techniques.
Fractional 57Fe absorption | Determined 2 weeks after iron intervention
  Fractional 57Fe absorption will be measured using stable-isotope techniques

CONTACTS AND LOCATIONS:
Overall Officials: Gary M. Brittenham, M.D., Principal Investigator — Columbia University
Locations (1):
- Hospital for Tropical Diseases, Mahidol University, Bangkok, Thailand